CLINICAL TRIAL: NCT02306382
Title: Randomized Controlled Multicenter Study for Diagnosis and Treatment of Perianal Abscesses.
Brief Title: Multicenter Study for Diagnosis and Treatment of Perianal Abscesses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Umeå (Other)
Responsible Party: Principal Investigator, Karin Gustafsson, MD, University Hospital, Umeå
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Gustafsson
Record Dates: First submitted 2012-12-13; First posted 2014-12-03 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Perianal Abscess; Anal Fistulas; Incontinence
Keywords: endoanal ultrasonography; drainage; perianal abscess; fistulas; incontience
MeSH Terms: conditions — Rectal Fistula; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ultrasonography, abscess (Experimental): The experimental group will be treated after examination with 3D ultrasonography. Follow up after two months and one year.
  Interventions: Procedure: Perianal abscess drainage; Device: 3D ultrasonography
- Control group with clincial inscision (Other): The control group will have drainage of their perianal abscess in the OR without ultrasound. Follow-up after two months and one year.
  Interventions: Procedure: Perianal abscess drainage

INTERVENTIONS:
Procedure: Perianal abscess drainage — The patientens will be randomly selected and after they have taken part and said yes to the study, half the group will undergo examination with ultrasound and half without. After this random selection all the patients abscess will be drained.
  Other Names: 1
Device: 3D ultrasonography — The patientens will be randomly selected and after they have taken part and said yes to the study, half the group will undergo examination with ultrasound and half without. After this random selection all the patients abscess will be drained.
  Other Names: 2
  Arms: ultrasonography, abscess

SUMMARY:
Drainage of perianal abscesses is a well established treatment. Traditionally its been done in general anesthesia after the swelling has been localised its been drained with a knife. After surgical intervention complications can occur with recidivism, chronic fistulas that go from the anal to the skin and sometimes the anal sphincter is damaged which can cause problems with incontinence.

Through ultrasound the abscess is opened under more controlled forms with a better visual overview. This is a new technique that has not been tested in larger studies. The aim with ultrasound-drainage as with traditional incision to drain the abscess so that the infected area can heal.

The hypothesis is a reduction of recurrences and formation of fistulas with the use of 3D ultrasonography.

DETAILED DESCRIPTION:
The individual patient is informed about the condition and if meets criteria is offered to take part in the study. Written information and informed consent always noted. Questions about the patients general medical condition is noted and if the person has had problems with perianal abscesses before.

ELIGIBILITY:
Inclusion Criteria:

* perianal abscess that needs surgical treatment, over the age of 18

Exclusion Criteria:

* Under the age of 18 or unable to understand study information because of language difficulties or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
adverse events | up to one year
  Patients will be assessed in the outpatient clinic after 2 months and 1 year after surgical treatment. Eventual complications may include anal sepsis, recurrence of anal abscess and fistula formation.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Gustafsson, MD, Principal Investigator — University Hospital, Umeå; Karin Strigård Strigård, MD, Study Director — University Hospital, Umeå; Ulf Gunnarsson, MD, Study Chair — University Hospital, Umeå
Locations (1):
- Department of Surgery, Umeå, County of Vasterbotten §, Sweden